CLINICAL TRIAL: NCT03776981
Title: The Effects of Core Activation and Stabilization Training on Gait Kinetics, Kinematics, and Speed, and Self-Perceived Function in Patients With Knee Osteoarthritis
Brief Title: Core Activation and Stabilization for Knee OA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Collaborators: Texas Woman's University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00001065; Study #20344 (Other: Texas Woman's University Institutional Review Board)
Record Dates: First submitted 2018-12-12; First posted 2018-12-17 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Osteoarthritis, Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Baseline Gait Comparisons of Groups (No Intervention): Determine if kinetic (time to first peak ground reaction force [T1] and second peak ground reaction force [F2], both in the sagittal plane) and kinematic (peak stance knee flexion angle [KFA] and external knee adduction moment [KAM]) gait variables, and speed, differ between patients with KOA and age and gender matched controls during self-selected paced ambulation, and determine which ones have predictive relationships with Knee Injury and Osteoarthritis Outcome Score (KOOS) scores in the patients with KOA.
- Gait with core activation (Experimental): Determine if volitional core activation alters gait kinetics (T1 and F2), kinematics (KFA and KAM), and speed in patients with and without KOA during self-selected paced ambulation when compared to ambulating without volitional core activation, and whether the subjective pain complaints are significantly changed in the group with KOA. Determine whether there are baseline differences in core activation between those with and without KOA.
  Interventions: Other: Core Activation
- Knee OA Gait After core stabilization (Experimental): Determine if a six-week core stabilization program alters KOOS score, and the kinetics (T1 and F2), kinematics (KFA and KAM), and speed of gait in patients with KOA during self-selected paced ambulation as compared to their pre-intervention baselines. Determine if there is a predictive relationship between the number of completed intervention sessions performed and these observed changes.
  Interventions: Other: Core Stabilization

INTERVENTIONS:
Other: Core Activation — Volitional activation of the transversus abdominis muscle during self-selected paced ambulation for both groups.
  Arms: Gait with core activation
Other: Core Stabilization — Six-week core stabilization program for the group of participants with knee osteoarthritis.
  Arms: Knee OA Gait After core stabilization

SUMMARY:
This will be the second investigation by the PI and sub-investigator on this topic, following the promising results of a pilot study on a small sample size (N=5) completed last year. Whether or not core stabilization influences gait impairments in patients with KOA remains to be seen. Core stabilization has been shown to have positive effects, including increased stride velocity and scores on functional tests like the Functional Reach Test and Timed Up and Go, in older adults. Older adults were also shown to have high compliance with a core stability training program. A systematic review indicated that core training is important to consider when treating older individuals to improve functional use of the extremities, improving participation in activities of daily living, and as part of a fall prevention program. Additionally, it has been shown to benefit young, active individuals in preventing anterior cruciate ligament injury and greater duration of improved outcomes in patients with patellofemoral pain syndrome. Athletes with decreased core control have been shown to be at an increased risk of knee injury as well. One potential cause for this is the ability of the core to improve lower extremity kinematics when activated during challenging single leg weight bearing activity. A recent publication by Azuma, et al. did indicate that paraspinal and anterior abdominal thinning had a negative predictive relationship to the presence of KOA; however, no investigation has explored a cause and effect relationship between core stability/stabilization training and the presence or severity of KOA, nor the gait and functional ability of patients with KOA. This later concept is the focus of this investigation.

DETAILED DESCRIPTION:
Unpublished pilot data collected by the same PI and sub-investigator shows that volitional activation of the TA during self-selected paced ambulation significantly decreases the time to first peak ground reaction force (T1) in the sagittal plane in participants with KOA (D.W. Flowers, C. Frilot, unpublished data, May 2018). This same kinetic gait variable is included in this investigation as one of the dependent variables in all three parts of the investigation.

Nearly four percent of the global population has KOA, with the global female percentage nearing five percent. Additionally, the years lived with disability (YLDs) resulting from the disorder increased by 64.8% from 1990 to 2010. The picture is not much better in the United States, where osteoarthritis ranks eighth highest in YLDs compared to other pathologies. The rate of KOA has continued to climb here in the U.S., doubling in the past half-century even when accounting for increased life expectancy and higher average BMI, both of which are considered risk factors in the development of KOA.

Patients with KOA have been shown to have gait abnormalities when compared to healthy controls, including alterations in trunk and pelvic kinematics, lower extremity kinematics and kinetics, gait speed, and functional outcome measure scores. Some of these differences, like an increased external knee adduction moment (KAM) and a decreased peak stance knee flexion angle (KFA), have been shown to correlate with the advancement of KOA and may be causative in nature. Others, like an increased T1 and reduced freely chosen gait speed, may be compensatory. The same has been found in regard to the reduced second peak ground reaction force in the sagittal plane (F2) observed in this population.

Reduced gait speed alone is predictive of increased fall risk in older adults, without any need to consider additional activities performed during walking tasks. Additionally, the gait impairments observed in this population can be so extreme that they can be more limiting than those observed in patients with diagnoses typically considered more severe, like congestive heart failure, diabetes, heart disease, and stroke. Therefore, improving function via improving gait speed via novel approaches is indicated, but not at the expense of increasing wear and tear on osteoarthritic joints. This investigation aims to show that core stabilization, which has been shown beneficially influence the kinetics and kinematics of lower extremity movements in younger, more active populations, can serve the same purpose in a population with KOA. The investigators are specifically trying to improve self-perceived function and gait speed, via improving the kinetics and kinematics observed in self-selected ambulation.

This investigation will be divided into three parts, each associated with one of the specific aims detailed in Section 1. All procedures will be performed in the School of Allied Health Professions, either in the Motion Analysis Laboratory (Gait Lab) or the Rehabilitation Faculty Practice (RFP) Clinic.

Part 1: Compare age and gender matched healthy controls and KOA groups on kinetics, kinematics, and gait speed during self-selected speed via a between groups analysis across the dependent variables, and determine if those differences in the KOA group have a predictive relationship with their KOOS scores.

Part 2: Within-group comparison of both groups (with and without volitional TA activation) and between-groups (control group versus KOA group). Compare pain levels during both conditions via VAS for the KOA group. Participants will wear biofeedback under both conditions, and all condition trials will be randomized. Alarm or verbal cue will be provided at 30% MVIC, and two electrodes placed over TA/obliquus internus (OI) just medial to anterior superior iliac spine (ASIS). A comparison of TA activation will be performed both within and between groups.

Part 3: Within-groups comparison of KOA group (pre-treatment and post-treatment; six-week training program) on kinetics, kinematics, and gait speed during self-selected paced ambulation. A comparison of KOOS scores before and after treatment with be performed as well.

Once recruitment and informed consent are completed:

Part 1: All participants will undergo anthropometric data collection first, including weight, height, leg length, knee joint width, and ankle joint width. Age matching will be done within +/- 5 years between the two groups. Reflective markers will then be placed on bilateral lower extremities following the Plug in Gait Model. EMG electrodes will be placed bilaterally just medial to the ASIS, over the TA/OI. The Gait Lab will undergo calibration, and the participant will undergo a static trial. In participants with bilateral KOA, the most painful limb, identified by subjective report, will be used in the data collection procedures. Healthy controls will undergo analysis of their dominant limb by indicating with which leg they would kick a ball.

Once the set-up and calibration are completed, the data collection will begin. The participant will be allowed a brief warm-up of 1-2 minutes, walking in the Gait Lab prior to data collection commences. The participant will then be asked to walk at a self-selected pace across the capture area until three trials with good force plate contact are obtained. Good force plate contact is defined as initial contact at the heel and pre-swing/toe off occurring on the force plate, and the absence of any evidence of distraction via the video cameras, such as the participant talking or looking around the lab. These three trials will be used in the kinetic, kinematic, and gait speed data analysis.

See Part 2 for additional trials that will be performed concurrently for both groups. Participants in the experimental group will also be asked to complete a KOOS questionnaire at the same time.

Part 2: Participants will undergo the same procedures described in Part 1 above. While the three trials are obtained for Part 1, three additional walking trials will be concurrently collected for the both groups. These will include the participant volitionally activating their TA during the walking trials, performed and screened exactly the same as in Part 1. These trials will be performed with and without audible biofeedback (via an alarm or verbal cueing), indicating the TA meeting the threshold subsequently discussed below. Investigators will randomly determine whether the trials with or without volitional TA activation are performed first (i.e., Part 1 versus Part 2 trials). The randomization done for Part 2 to determine whether or not the without (Part 1) or with (Part 2) volitional TA activation trials are performed first will be determined via random number generation between 0 and 1 in Excel. Those with 0 will perform the without volitional TA (Part 1) trials first, while those with 1 will perform the with volitional TA activation trials (Part 2) first.

The patient will lie supine on the mat in the lab and will be taught how to perform a TA contraction. Please see the attached script with the instructions that will be used in this education. A baseline maximal contraction will be performed supine, and the amplitude of contraction will be considered maximal voluntary isometric contraction (MVIC). The device will be set to provide audible feedback, or the participant will receive a verbal cue from the investigator, at 30% MVIC. This feedback will be randomized throughout the trials with TA activation via random number generation in Excel, with 0 signifying no cue and 1 indicating a cue. The task will be repeated seated, then standing, prior to data collection.

The experimental group, during both sets of trials, will be asked to subjectively rate their perceived pain in the lower extremity being used in data collection via a 10-point scale, typically used on the VAS, although no visual will be used. Please see the supplemental script document attached to this protocol for the instructions used.

Part 3: Participants in the experimental group will participate in a six-week core stabilization intervention program. Please see the attached intervention program. This program will commence as soon as possible after Parts 1 and 2 of the investigation are completed. Participants will participate in two scheduled intervention sessions each week. Additionally, there will be a home exercise program, consisting of exercises from each week to be performed at home independently. Participants will be provided education and a handout on these exercises by the PI, which will include directions, photographs of the exercises, and a completion check-off for each session. These will be performed three times per week, every other day. The PI will be coordinator of the scheduling and performance of these interventions. These intervention sessions will be performed in the RFP Clinic in the SAHP, either in the open gym or in a private treatment room. This decision will be left up to the participant. More than one participant may or may not undergo intervention with the PI simultaneously, but only with the participants' consent. No more than three participants will undergo the training simultaneously. Training sessions will not be performed on consecutive days in an effort to reduce the chances of delayed onset muscle soreness being present during treatment sessions. Additionally, the core training program includes predetermined guidelines on exercise progressions in order to ensure that the exercises are not progressed too rapidly. The PI will be present and will lead all sessions, ensuring that the exercises and their progressions are done correctly.

After the completion of the intervention program, each participant will undergo gait analysis in the same manner mentioned in Part 1, with the exception of no anthropometric data being collected. Participants will then complete a second, post-intervention KOOS questionnaire, and turn in their home exercise program sheet with tallies from completed sessions. Please see Part 1 for completion of the pre-intervention KOOS questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking men and women
* 40 years old and older
* any race or ethnic group
* a documented diagnosis from a medical provider (i.e., physician, physician assistant, or nurse practitioner, etc.) of KOA, unilaterally or bilaterally.
* Previous or current physical therapy patients may be included (see exclusion criteria for exceptions).

Healthy controls will meet the same requirements, but:

* without a medical diagnosis of KOA
* have the ability to ambulate on a level surface without any report of pain in their knees at the time of gait assessment.

Exclusion Criteria:

* Those with other lower extremity injuries (orthopaedic, cardiovascular, neurologic, etc.) which are currently hindering their ability to ambulate
* those with current complaints of low back pain
* those who have undergone bilateral total knee arthroplasty
* those with concomitant diagnosis of rheumatoid arthritis
* those persons not able to ambulate independently with or without an assistive device
* those who have received a corticosteroid injection within the past two months
* those who have received a hyaluronic acid injection in the past six months
* those persons currently enrolled in a core training program as part of formal physical therapy or physical fitness.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-01-08 (Actual); Primary Completion 2019-12-11 (Actual); Study Completion 2019-12-11 (Actual)

PRIMARY OUTCOMES:
Time to First Peak Ground Reaction Force in the Sagittal Plane (T1) | Through study completion, on average about 1 year.
  Kinetic variable observed during gait analysis.
Second Peak Ground Reaction Force in the Sagittal Plane (F2) | Through study completion, on average about 1 year.
  Kinetic variable observed during gait analysis.
Peak Stance Knee Flexion Angle (KFA) | Through study completion, on average about 1 year.
  Kinematic variable observed during gait analysis.
External Knee Adduction Moment (KAM) | Through study completion, on average about 1 year.
  Kinematic variable observed during gait analysis.
Gait Speed | Through study completion, on average about 1 year.
  Self-selected gait velocity of each participant during gait analysis.

SECONDARY OUTCOMES:
Pain Rating on Visual Analog Scale (VAS) | Through study completion, on average about 1 year.
  Self-perceived rating of pain related by participants.
Knee Injury and Osteoarthritis Outcome Score (KOOS) | Through study completion, on average about 1 year.
  Outcome measure for self-perceived function in patients with knee osteoarthritis.
Transversus Abdominis Activation | Through study completion, on average about 1 year.
  Transversus abdominis activity as measured via electromyography.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel W Flowers, DPT, Principal Investigator — Louisiana State University Health Sciences Center Shreveport
Locations (1):
- Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Granacher U, Lacroix A, Muehlbauer T, Roettger K, Gollhofer A. Effects of core instability strength training on trunk muscle strength, spinal mobility, dynamic balance and functional mobility in older adults. Gerontology. 2013;59(2):105-13. doi: 10.1159/000343152. Epub 2012 Oct 24. PMID 23108436
- [Background] Granacher U, Gollhofer A, Hortobagyi T, Kressig RW, Muehlbauer T. The importance of trunk muscle strength for balance, functional performance, and fall prevention in seniors: a systematic review. Sports Med. 2013 Jul;43(7):627-41. doi: 10.1007/s40279-013-0041-1. PMID 23568373
- [Background] Whyte EF, Richter C, O'Connor S, Moran KA. Effects of a dynamic core stability program on the biomechanics of cutting maneuvers: A randomized controlled trial. Scand J Med Sci Sports. 2018 Feb;28(2):452-462. doi: 10.1111/sms.12931. Epub 2017 Jul 13. PMID 28605148
- [Background] Ferber R, Bolgla L, Earl-Boehm JE, Emery C, Hamstra-Wright K. Strengthening of the hip and core versus knee muscles for the treatment of patellofemoral pain: a multicenter randomized controlled trial. J Athl Train. 2015 Apr;50(4):366-77. doi: 10.4085/1062-6050-49.3.70. Epub 2014 Nov 3. PMID 25365133
- [Background] Zazulak BT, Hewett TE, Reeves NP, Goldberg B, Cholewicki J. Deficits in neuromuscular control of the trunk predict knee injury risk: a prospective biomechanical-epidemiologic study. Am J Sports Med. 2007 Jul;35(7):1123-30. doi: 10.1177/0363546507301585. Epub 2007 Apr 27. PMID 17468378
- [Background] Shirey M, Hurlbutt M, Johansen N, King GW, Wilkinson SG, Hoover DL. The influence of core musculature engagement on hip and knee kinematics in women during a single leg squat. Int J Sports Phys Ther. 2012 Feb;7(1):1-12. PMID 22319676
- [Background] Azuma K, Sera Y, Shinjo T, Takayama M, Shiomi E, Momoshima S, Iwao Y, Ishida H, Matsumoto H. Maintenance of the paraspinal muscles may protect against radiographic knee osteoarthritis. Open Access Rheumatol. 2017 Aug 10;9:151-158. doi: 10.2147/OARRR.S130688. eCollection 2017. PMID 28860877
- [Background] Vos T, Flaxman AD, Naghavi M, Lozano R, Michaud C, Ezzati M, Shibuya K, Salomon JA, Abdalla S, Aboyans V, Abraham J, Ackerman I, Aggarwal R, Ahn SY, Ali MK, Alvarado M, Anderson HR, Anderson LM, Andrews KG, Atkinson C, Baddour LM, Bahalim AN, Barker-Collo S, Barrero LH, Bartels DH, Basanez MG, Baxter A, Bell ML, Benjamin EJ, Bennett D, Bernabe E, Bhalla K, Bhandari B, Bikbov B, Bin Abdulhak A, Birbeck G, Black JA, Blencowe H, Blore JD, Blyth F, Bolliger I, Bonaventure A, Boufous S, Bourne R, Boussinesq M, Braithwaite T, Brayne C, Bridgett L, Brooker S, Brooks P, Brugha TS, Bryan-Hancock C, Bucello C, Buchbinder R, Buckle G, Budke CM, Burch M, Burney P, Burstein R, Calabria B, Campbell B, Canter CE, Carabin H, Carapetis J, Carmona L, Cella C, Charlson F, Chen H, Cheng AT, Chou D, Chugh SS, Coffeng LE, Colan SD, Colquhoun S, Colson KE, Condon J, Connor MD, Cooper LT, Corriere M, Cortinovis M, de Vaccaro KC, Couser W, Cowie BC, Criqui MH, Cross M, Dabhadkar KC, Dahiya M, Dahodwala N, Damsere-Derry J, Danaei G, Davis A, De Leo D, Degenhardt L, Dellavalle R, Delossantos A, Denenberg J, Derrett S, Des Jarlais DC, Dharmaratne SD, Dherani M, Diaz-Torne C, Dolk H, Dorsey ER, Driscoll T, Duber H, Ebel B, Edmond K, Elbaz A, Ali SE, Erskine H, Erwin PJ, Espindola P, Ewoigbokhan SE, Farzadfar F, Feigin V, Felson DT, Ferrari A, Ferri CP, Fevre EM, Finucane MM, Flaxman S, Flood L, Foreman K, Forouzanfar MH, Fowkes FG, Franklin R, Fransen M, Freeman MK, Gabbe BJ, Gabriel SE, Gakidou E, Ganatra HA, Garcia B, Gaspari F, Gillum RF, Gmel G, Gosselin R, Grainger R, Groeger J, Guillemin F, Gunnell D, Gupta R, Haagsma J, Hagan H, Halasa YA, Hall W, Haring D, Haro JM, Harrison JE, Havmoeller R, Hay RJ, Higashi H, Hill C, Hoen B, Hoffman H, Hotez PJ, Hoy D, Huang JJ, Ibeanusi SE, Jacobsen KH, James SL, Jarvis D, Jasrasaria R, Jayaraman S, Johns N, Jonas JB, Karthikeyan G, Kassebaum N, Kawakami N, Keren A, Khoo JP, King CH, Knowlton LM, Kobusingye O, Koranteng A, Krishnamurthi R, Lalloo R, Laslett LL, Lathlean T, Leasher JL, Lee YY, Leigh J, Lim SS, Limb E, Lin JK, Lipnick M, Lipshultz SE, Liu W, Loane M, Ohno SL, Lyons R, Ma J, Mabweijano J, MacIntyre MF, Malekzadeh R, Mallinger L, Manivannan S, Marcenes W, March L, Margolis DJ, Marks GB, Marks R, Matsumori A, Matzopoulos R, Mayosi BM, McAnulty JH, McDermott MM, McGill N, McGrath J, Medina-Mora ME, Meltzer M, Mensah GA, Merriman TR, Meyer AC, Miglioli V, Miller M, Miller TR, Mitchell PB, Mocumbi AO, Moffitt TE, Mokdad AA, Monasta L, Montico M, Moradi-Lakeh M, Moran A, Morawska L, Mori R, Murdoch ME, Mwaniki MK, Naidoo K, Nair MN, Naldi L, Narayan KM, Nelson PK, Nelson RG, Nevitt MC, Newton CR, Nolte S, Norman P, Norman R, O'Donnell M, O'Hanlon S, Olives C, Omer SB, Ortblad K, Osborne R, Ozgediz D, Page A, Pahari B, Pandian JD, Rivero AP, Patten SB, Pearce N, Padilla RP, Perez-Ruiz F, Perico N, Pesudovs K, Phillips D, Phillips MR, Pierce K, Pion S, Polanczyk GV, Polinder S, Pope CA 3rd, Popova S, Porrini E, Pourmalek F, Prince M, Pullan RL, Ramaiah KD, Ranganathan D, Razavi H, Regan M, Rehm JT, Rein DB, Remuzzi G, Richardson K, Rivara FP, Roberts T, Robinson C, De Leon FR, Ronfani L, Room R, Rosenfeld LC, Rushton L, Sacco RL, Saha S, Sampson U, Sanchez-Riera L, Sanman E, Schwebel DC, Scott JG, Segui-Gomez M, Shahraz S, Shepard DS, Shin H, Shivakoti R, Singh D, Singh GM, Singh JA, Singleton J, Sleet DA, Sliwa K, Smith E, Smith JL, Stapelberg NJ, Steer A, Steiner T, Stolk WA, Stovner LJ, Sudfeld C, Syed S, Tamburlini G, Tavakkoli M, Taylor HR, Taylor JA, Taylor WJ, Thomas B, Thomson WM, Thurston GD, Tleyjeh IM, Tonelli M, Towbin JA, Truelsen T, Tsilimbaris MK, Ubeda C, Undurraga EA, van der Werf MJ, van Os J, Vavilala MS, Venketasubramanian N, Wang M, Wang W, Watt K, Weatherall DJ, Weinstock MA, Weintraub R, Weisskopf MG, Weissman MM, White RA, Whiteford H, Wiersma ST, Wilkinson JD, Williams HC, Williams SR, Witt E, Wolfe F, Woolf AD, Wulf S, Yeh PH, Zaidi AK, Zheng ZJ, Zonies D, Lopez AD, Murray CJ, AlMazroa MA, Memish ZA. Years lived with disability (YLDs) for 1160 sequelae of 289 diseases and injuries 1990-2010: a systematic analysis for the Global Burden of Disease Study 2010. Lancet. 2012 Dec 15;380(9859):2163-96. doi: 10.1016/S0140-6736(12)61729-2. PMID 23245607
- [Background] Murray CJ, Atkinson C, Bhalla K, Birbeck G, Burstein R, Chou D, Dellavalle R, Danaei G, Ezzati M, Fahimi A, Flaxman D, Foreman, Gabriel S, Gakidou E, Kassebaum N, Khatibzadeh S, Lim S, Lipshultz SE, London S, Lopez, MacIntyre MF, Mokdad AH, Moran A, Moran AE, Mozaffarian D, Murphy T, Naghavi M, Pope C, Roberts T, Salomon J, Schwebel DC, Shahraz S, Sleet DA, Murray, Abraham J, Ali MK, Atkinson C, Bartels DH, Bhalla K, Birbeck G, Burstein R, Chen H, Criqui MH, Dahodwala, Jarlais, Ding EL, Dorsey ER, Ebel BE, Ezzati M, Fahami, Flaxman S, Flaxman AD, Gonzalez-Medina D, Grant B, Hagan H, Hoffman H, Kassebaum N, Khatibzadeh S, Leasher JL, Lin J, Lipshultz SE, Lozano R, Lu Y, Mallinger L, McDermott MM, Micha R, Miller TR, Mokdad AA, Mokdad AH, Mozaffarian D, Naghavi M, Narayan KM, Omer SB, Pelizzari PM, Phillips D, Ranganathan D, Rivara FP, Roberts T, Sampson U, Sanman E, Sapkota A, Schwebel DC, Sharaz S, Shivakoti R, Singh GM, Singh D, Tavakkoli M, Towbin JA, Wilkinson JD, Zabetian A, Murray, Abraham J, Ali MK, Alvardo M, Atkinson C, Baddour LM, Benjamin EJ, Bhalla K, Birbeck G, Bolliger I, Burstein R, Carnahan E, Chou D, Chugh SS, Cohen A, Colson KE, Cooper LT, Couser W, Criqui MH, Dabhadkar KC, Dellavalle RP, Jarlais, Dicker D, Dorsey ER, Duber H, Ebel BE, Engell RE, Ezzati M, Felson DT, Finucane MM, Flaxman S, Flaxman AD, Fleming T, Foreman, Forouzanfar MH, Freedman G, Freeman MK, Gakidou E, Gillum RF, Gonzalez-Medina D, Gosselin R, Gutierrez HR, Hagan H, Havmoeller R, Hoffman H, Jacobsen KH, James SL, Jasrasaria R, Jayarman S, Johns N, Kassebaum N, Khatibzadeh S, Lan Q, Leasher JL, Lim S, Lipshultz SE, London S, Lopez, Lozano R, Lu Y, Mallinger L, Meltzer M, Mensah GA, Michaud C, Miller TR, Mock C, Moffitt TE, Mokdad AA, Mokdad AH, Moran A, Naghavi M, Narayan KM, Nelson RG, Olives C, Omer SB, Ortblad K, Ostro B, Pelizzari PM, Phillips D, Raju M, Razavi H, Ritz B, Roberts T, Sacco RL, Salomon J, Sampson U, Schwebel DC, Shahraz S, Shibuya K, Silberberg D, Singh JA, Steenland K, Taylor JA, Thurston GD, Vavilala MS, Vos T, Wagner GR, Weinstock MA, Weisskopf MG, Wulf S, Murray; U.S. Burden of Disease Collaborators. The state of US health, 1990-2010: burden of diseases, injuries, and risk factors. JAMA. 2013 Aug 14;310(6):591-608. doi: 10.1001/jama.2013.13805. PMID 23842577
- [Background] Wallace IJ, Worthington S, Felson DT, Jurmain RD, Wren KT, Maijanen H, Woods RJ, Lieberman DE. Knee osteoarthritis has doubled in prevalence since the mid-20th century. Proc Natl Acad Sci U S A. 2017 Aug 29;114(35):9332-9336. doi: 10.1073/pnas.1703856114. Epub 2017 Aug 14. PMID 28808025
- [Background] Felson DT, Lawrence RC, Dieppe PA, Hirsch R, Helmick CG, Jordan JM, Kington RS, Lane NE, Nevitt MC, Zhang Y, Sowers M, McAlindon T, Spector TD, Poole AR, Yanovski SZ, Ateshian G, Sharma L, Buckwalter JA, Brandt KD, Fries JF. Osteoarthritis: new insights. Part 1: the disease and its risk factors. Ann Intern Med. 2000 Oct 17;133(8):635-46. doi: 10.7326/0003-4819-133-8-200010170-00016. PMID 11033593
- [Background] Linley HS, Sled EA, Culham EG, Deluzio KJ. A biomechanical analysis of trunk and pelvis motion during gait in subjects with knee osteoarthritis compared to control subjects. Clin Biomech (Bristol). 2010 Dec;25(10):1003-10. doi: 10.1016/j.clinbiomech.2010.07.012. Epub 2010 Sep 6. PMID 20822836
- [Background] Al-Zahrani KS, Bakheit AM. A study of the gait characteristics of patients with chronic osteoarthritis of the knee. Disabil Rehabil. 2002 Mar 20;24(5):275-80. doi: 10.1080/09638280110087098. PMID 12004973
- [Background] Astephen JL, Deluzio KJ, Caldwell GE, Dunbar MJ. Biomechanical changes at the hip, knee, and ankle joints during gait are associated with knee osteoarthritis severity. J Orthop Res. 2008 Mar;26(3):332-41. doi: 10.1002/jor.20496. PMID 17960658
- [Background] Kumar D, Manal KT, Rudolph KS. Knee joint loading during gait in healthy controls and individuals with knee osteoarthritis. Osteoarthritis Cartilage. 2013 Feb;21(2):298-305. doi: 10.1016/j.joca.2012.11.008. Epub 2012 Nov 24. PMID 23182814
- [Background] Chen CP, Chen MJ, Pei YC, Lew HL, Wong PY, Tang SF. Sagittal plane loading response during gait in different age groups and in people with knee osteoarthritis. Am J Phys Med Rehabil. 2003 Apr;82(4):307-12. doi: 10.1097/01.PHM.0000056987.33630.56. PMID 12649658
- [Background] Duffell LD, Jordan SJ, Cobb JP, McGregor AH. Gait adaptations with aging in healthy participants and people with knee-joint osteoarthritis. Gait Posture. 2017 Sep;57:246-251. doi: 10.1016/j.gaitpost.2017.06.015. Epub 2017 Jun 21. PMID 28672154
- [Background] Messier SP, Loeser RF, Hoover JL, Semble EL, Wise CM. Osteoarthritis of the knee: effects on gait, strength, and flexibility. Arch Phys Med Rehabil. 1992 Jan;73(1):29-36. PMID 1729969
- [Background] Huang SC, Wei IP, Chien HL, Wang TM, Liu YH, Chen HL, Lu TW, Lin JG. Effects of severity of degeneration on gait patterns in patients with medial knee osteoarthritis. Med Eng Phys. 2008 Oct;30(8):997-1003. doi: 10.1016/j.medengphy.2008.02.006. Epub 2008 Apr 15. PMID 18417411
- [Background] Zeni JA Jr, Higginson JS. Differences in gait parameters between healthy subjects and persons with moderate and severe knee osteoarthritis: a result of altered walking speed? Clin Biomech (Bristol). 2009 May;24(4):372-8. doi: 10.1016/j.clinbiomech.2009.02.001. Epub 2009 Mar 13. PMID 19285768
- [Background] Miyazaki T, Wada M, Kawahara H, Sato M, Baba H, Shimada S. Dynamic load at baseline can predict radiographic disease progression in medial compartment knee osteoarthritis. Ann Rheum Dis. 2002 Jul;61(7):617-22. doi: 10.1136/ard.61.7.617. PMID 12079903
- [Background] Favre J, Erhart-Hledik JC, Chehab EF, Andriacchi TP. Baseline ambulatory knee kinematics are associated with changes in cartilage thickness in osteoarthritic patients over 5 years. J Biomech. 2016 Jun 14;49(9):1859-1864. doi: 10.1016/j.jbiomech.2016.04.029. Epub 2016 Apr 29. PMID 27178021
- [Background] Messier SP. Osteoarthritis of the knee and associated factors of age and obesity: effects on gait. Med Sci Sports Exerc. 1994 Dec;26(12):1446-52. PMID 7869877
- [Background] Menant JC, Schoene D, Sarofim M, Lord SR. Single and dual task tests of gait speed are equivalent in the prediction of falls in older people: a systematic review and meta-analysis. Ageing Res Rev. 2014 Jul;16:83-104. doi: 10.1016/j.arr.2014.06.001. Epub 2014 Jun 7. PMID 24915643
- [Background] Guccione AA, Felson DT, Anderson JJ, Anthony JM, Zhang Y, Wilson PW, Kelly-Hayes M, Wolf PA, Kreger BE, Kannel WB. The effects of specific medical conditions on the functional limitations of elders in the Framingham Study. Am J Public Health. 1994 Mar;84(3):351-8. doi: 10.2105/ajph.84.3.351. PMID 8129049
- [Background] Shi H, Huang H, Yu Y, Liang Z, Zhang S, Yu B, Liu H, Ao Y. Effect of dual task on gait asymmetry in patients after anterior cruciate ligament reconstruction. Sci Rep. 2018 Aug 13;8(1):12057. doi: 10.1038/s41598-018-30459-w. PMID 30104568
- [Background] Tang SF, Chen CP, Chen MJ, Pei YC, Lau YC, Leong CP. Changes in sagittal ground reaction forces after intra-articular hyaluronate injections for knee osteoarthritis. Arch Phys Med Rehabil. 2004 Jun;85(6):951-5. doi: 10.1016/j.apmr.2003.08.095. PMID 15179649
- [Background] Rue JP, Yanke AB, Busam ML, McNickle AG, Cole BJ. Prospective evaluation of concurrent meniscus transplantation and articular cartilage repair: minimum 2-year follow-up. Am J Sports Med. 2008 Sep;36(9):1770-8. doi: 10.1177/0363546508317122. Epub 2008 May 15. PMID 18483199
- [Derived] Flowers DW, Brewer W, Ellison J, Mitchell K, Frilot C. Transversus abdominis activation does not alter gait impairments in patients with and without knee osteoarthritis. Clin Biomech (Bristol). 2021 Feb;82:105270. doi: 10.1016/j.clinbiomech.2020.105270. Epub 2021 Jan 1. PMID 33421757

DOCUMENTS (2):
  • Informed Consent Form (2018-11-08): https://cdn.clinicaltrials.gov/large-docs/81/NCT03776981/ICF_001.pdf
  • Study Protocol and Statistical Analysis Plan (2019-07-26): https://cdn.clinicaltrials.gov/large-docs/81/NCT03776981/Prot_SAP_003.pdf